CLINICAL TRIAL: NCT04175340
Title: A Safety and Effectiveness Study of a New Preservative Free Rewetting Drop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 952
Record Dates: First submitted 2019-11-20; First posted 2019-11-25 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2023-06

CONDITIONS: Contact Lens Wear

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BL-300-PFM04 (Experimental)
  Interventions: Device: BL-300-PFM04
- Lubricating and rewetting drops (Active Comparator)
  Interventions: Device: OPTI-FREE

INTERVENTIONS:
Device: BL-300-PFM04 — Preservative Free Lubricating and Rewetting Drops for use during contact lens wear
  Arms: BL-300-PFM04
Device: OPTI-FREE — Replenish Rewetting Drops
  Arms: Lubricating and rewetting drops

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of lubricating and rewetting drop (Test) compared to OPTI-FREE® Replenish® Rewetting Drops (Control) when used by habitual contact lens wearers to bilaterally lubricate and rewet soft (hydrophilic) contact lenses including silicone hydrogel contact lenses and gas permeable (silicone acrylate and fluoro silicone acrylate) contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be of legal age (at least 18) on the date the Informed Consent Form (ICF) is signed and have the capacity to provide voluntary informed consent
* Subjects must be habitual wearers of included contact lenses.
* Subjects must be adapted lens wearers and wear a lens in each eye and each lens must be of the same manufacture and brand.
* Subjects must agree to wear their lenses on a daily wear basis for approximately 1 month.

Exclusion Criteria:

• Subjects participating in any drug or device clinical investigation within two weeks prior to entry into this study and/or during the period of study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Bausch Site 108, San Francisco, California
  - Bausch Site 111, Torrance, California
  - Bausch Site 106, Sarasota, Florida
  - Bausch Site 104, Decatur, Georgia
  - Bausch Site 110, Bloomington, Kansas
  - Bausch Site 112, Leavenworth, Kansas
  - Bausch Site 107, Portland, Maine
  - Bausch Site 109, Edina, Minnesota
  - Bausch Site 102, Jamestown, New York
  - Bausch Site 113, Vestal, New York
  - Bausch Site 101, Miamisburg, Ohio
  - Bausch Site 105, West Chester, Ohio
  - Bausch Site 114, Grants Pass, Oregon
  - Bausch Site 115, Brentwood, Tennessee
  - Bausch Site 103, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | BL-300-PFM04 | Lubricating and Rewetting Drops
Started | 188; 376 Eyes | 181; 362 Eyes
Completed | 188; 376 Eyes | 181; 362 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BL-300-PFM04 | Lubricating and Rewetting Drops | Total
Number analyzed (Participants) | 188 | 181 | 369
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 188 | 181 | 369
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.6 (9.56) | 33.7 (8.57) | 34.6 (9.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 57 | 117
  Male | 128 | 124 | 252
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 24 | 27 | 51
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 18 | 21 | 39
  White | 144 | 130 | 274
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 188 | 181 | 369

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort Averaged Over All Follow-up Visits
Description: Overall comfort will be assessed for each eye on a scale from 0 to 100, with 100 denoting the most favorable response. For each eye, mean overall comfort over all follow-up visits will be computed as the average of the non-missing values overall scheduled follow-up visits.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | BL-300-PFM04 | Lubricating and Rewetting Drops
Number analyzed (Participants) | 184 | 177
Number analyzed (Eyes) | 368 | 354
units on a scale | 91.72 (9.988) | 91.54 (10.680)

2. Primary Outcome: Dryness Averaged Over All Follow-up Visits
Description: Dryness will be assessed for each eye on a scale from 0 to 100, with 100 denoting the most favorable response. For each eye, mean dryness over all follow-up visits will be computed as the average of the non-missing values over all scheduled follow-up visits.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | BL-300-PFM04 | Lubricating and Rewetting Drops
Number analyzed (Participants) | 184 | 177
Number analyzed (Eyes) | 368 | 354
units on a scale | 87.91 (13.332) | 87.01 (14.650)

3. Primary Outcome: Proportion of Eyes With Slit Lamp Findings Greater Than Grade 2 at Any Follow-up Visit
Description: At each follow-up visit, graded slit lamp findings will be assessed for each eye using Grades 0 through 4. Using only the non-missing observations from all visits without imputation, each eye will be classified with respect to findings greater than grade 2 at any visit (Absent, Present).
Time Frame: 1 month
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | BL-300-PFM04 | Lubricating and Rewetting Drops
Number analyzed (Participants) | 187 | 180
Number analyzed (Eyes) | 374 | 360
Eyes | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 Month
Arm/Group | BL-300-PFM04 | Lubricating and Rewetting Drops
All-Cause Mortality (participants affected / at risk) | 0/188 | 0/181
Serious Adverse Events (participants affected / at risk) | 0/188 | 0/181
Other Adverse Events (participants affected / at risk) | 0/188 | 0/181

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT04175340/Prot_SAP_000.pdf